CLINICAL TRIAL: NCT06153407
Title: Genetic Test Based Risk Prediction of Early Calcific Aortic Valve Disease in Patients With Bicuspid Aortic Valve
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2023-1045
Record Dates: First submitted 2023-11-10; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Bicuspid Aortic Valve
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to elucidate the impact of germline mutations and clonal hematopoiesis (CHIP) on the progression of early aortic valve calcification in patients with bicuspid aortic valves. The study will be conducted over a recruitment period of one year and a follow-up observation period of two years. Considering a 2-year event rate and a 33% occurrence rate of clonal hematopoiesis, each group requires a minimum of 102 participants. Accounting for a 15% dropout rate, a total of 120 participants are needed for each group (type I error (α) = 5%, type II error (β) = 20%). Therefore, the total study population, including patients with normal aortic valve function, is set at 240 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed bicuspid aortic valves based on cardiac imaging (echocardiography, CT, MRI) or surgical findings.
2. Early aortic valve calcification group: Patients aged 20-80 with moderate or greater aortic valve stenosis/regurgitation.
3. Normal functioning aortic valve group: Patients aged 20-80 with mild or less aortic valve stenosis/regurgitation.
4. Patients who understand the purpose of the study and voluntarily consent to participate.

Exclusion Criteria:

1. Patients with malignant neoplastic diseases or other conditions, such as cerebrovascular accidents, which predict survival of less than 6 months.
2. Patients with unclear presence of bicuspid aortic valves.
3. Patients with stage 3 or higher chronic kidney disease.
4. Patients with other inherited cardiac conditions.
5. Patients with cognitive impairment or hemodynamically unstable patients who have difficulty understanding the study content.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who have bicuspid aortic valve
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Presence of germline mutation | 2 years follow-up
Clonal hematopoiesis of indeterminate potential (CHIP) mutation | 2 years follow-up
  Clonal hematopoiesis of indeterminate potential (CHIP) is the presence of a clonally expanded hematopoietic stem cell caused by a leukemogenic mutation.

SECONDARY OUTCOMES:
Progression of aortic valve calcification | 2 years follow-up
  Progression of aortic valve calcification measured by computed tomography (AV calcium score) or Echocardiography (Progression of AS/AR)

CONTACTS AND LOCATIONS:
Overall Officials: Iksung Cho, Principal Investigator — Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Division of Cardiology, Yonsei University Health System, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No